CLINICAL TRIAL: NCT05091281
Title: Macintosh Laryngoscope Versus GlideScope® Versus C-MAC®(D) Videolaryngoscope for Double Lumen Endotracheal Intubation in Patients Undergoing Thoracic Surgery
Brief Title: Macintosh Versus GlideScope Versus C-MAC for Double Lumen Endotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Mogahed, Associate professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 34776/7/21
Record Dates: First submitted 2021-10-01; First posted 2021-10-25 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Thoracic
Keywords: Macintosh; laryngoscope; GlideScope; C-MAC; videolaryngoscope; double lumen tube

STUDY DESIGN:
Intervention Model Description: Patients randomly assigned into Macintosh group, GlideScope (Verathon Medical, Bothwell, UT, USA) group, or CMAC(D) (Karl Storz GmbHand Co.KG, Tuttlingen, Germany) group. After pre-oxygenation , anesthesia will be induced with intravenous midazolam 0.05 mg. kg- 1 , propofol 1.5 mg. kg- 1 , fentanyl 5 μg. kg- 1 , and rocuronium 0.6 mg. kg- 1 . . The DLT will be inserted with the distal concavity facing anteriorly until the bronchial lumen cuff passed the vocal cords. The stylet will be then removed, and rotation will be performed while tube will be advanced. The left DLT rotated 90° counter-clockwise, and the right DLT will be rotated 90° clockwise to enter the respective mainstem bronchus.
Who Masked: Participant
Masking Description: Before the study, the computerized randomization will be performed and the allocation results will be placed in individual numbered and sealed envelopes. Patients remained blinded about their intubation technique until post-operative assessment was completed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): After induction of anesthesia intubation was done by Macintosh laryngoscope
  Interventions: Device: Intubation of the double lumen tube by Macintoch laryngoscope
- Group II (Active Comparator): After induction of anesthesia intubation was done by GlideScope®videolaryngoscope
  Interventions: Device: Intubation of the double lumen tube by Glidescope videolaryngoscope
- Group III (Active Comparator): After induction of anesthesia intubation was done byC-MAC®(D) videolaryngoscope
  Interventions: Device: Intubation of the double lumen tube by C-MAC®(D) videolaryngoscope

INTERVENTIONS:
Device: Intubation of the double lumen tube by Macintoch laryngoscope — After induction of anesthesia insertion of the double lumen tube was done by Macintosh laryngoscope
  Arms: Group I
Device: Intubation of the double lumen tube by Glidescope videolaryngoscope — After induction of anesthesia insertion of the double lumen tube was done by GlideScope® videolaryngoscope
  Arms: Group II
Device: Intubation of the double lumen tube by C-MAC®(D) videolaryngoscope — After induction of anesthesia insertion of the double lumen tube was done by C-MAC®(D) videolaryngoscope
  Arms: Group III

SUMMARY:
The double lumen endotracheal tube (DLT) is the most widely-used device for single lung ventilation in current thoracic anesthesia practice. In recent years, the routine application of the videolaryngoscope for single lumen endotracheal intubation has increased; nevertheless there are few studies of the use of the videolaryngoscope for DLT. The authors wondered whether there were benefits to using the videolaryngoscope for DLT placement in patients with predicted normal airways. Therefore, this study was designed to compare the performances of the GlideScope®, the C-MAC®(D) videolaryngoscope and the Macintosh laryngoscope in DLT intubation.

DETAILED DESCRIPTION:
Patients randomly assigned into Macintosh group, GlideScope (Verathon Medical, Bothwell, UT, USA) group, or CMAC(D) (Karl Storz GmbHand Co.KG, Tuttlingen, Germany) group. This will be done using a closed envelope technique using a computer-generated block randomization method. Before the study, the computerized randomization will be performed and the allocation results will be placed in individual numbered and sealed envelopes. Patients remained blinded about their intubation technique until post-operative assessment was completed. The researcher responsible for recruitment will be blinded to the allocation result. After a patient will be consented for the study, allocation will be revealed. All endotracheal intubations will be performed by fthe same anesthesiologist with 10 years' working experience skilled in videolaryngoscopy. Left-side or right-side 32Fr/35Fr Mallinckrodt™ DLTs (Mallinckrodt Medical, Athlone, Ireland) will be selected for female patients and 35Fr/37Fr DLTs for male patients depending on whether their heights were below or above 155 cm for females and 165 cm for males. If the operation side will be the left, right-side DLT will be used; otherwise, the left-side DLT will be used. To facilitate intubation, the distal 10-12 cm concavity of the DLT (with the stylet in situ) will be molded along the blade convexity in each group. The tracheal and the bronchial cuffs of the DLT tubes will be lubricated with sterile Surgilube. No premedication will be given before induction. Standard monitoring prior to induction included ECG, invasive arterial blood pressure, SpO2, and end-tidal carbon dioxide. After pre-oxygenation with 100% oxygen, anesthesia will be induced with intravenous midazolam 0.05 mg. kg- 1 , propofol 1.5 mg. kg- 1 , fentanyl 5 μg. kg- 1 , and rocuronium 0.6 mg. kg- 1 . Two minutes after rocuronium administration, DLT intubation will be performed using the allocated laryngoscope. The DLT will be inserted with the distal concavity facing anteriorly until the bronchial lumen cuff passed the vocal cords. The stylet will be then removed, and rotation will be performed while tube will be advanced. The left DLT rotated 90° counter-clockwise, and the right DLT will be rotated 90° clockwise to enter the respective mainstem bronchus. The number of intubation attempts, ease of laryngoscopy insertion, Quality of view, Assist maneuvers, Intubation difficulty will be recorded. Hemodynamic changes will be monitored during induction. If systolic blood pressure fell below 80 mmHg, ephedrine 5 mg will be administrated intravenously. Atropine 0.5 mg will be given for heart rate below 50 beats per minute. After the tip of the DLT was located in the targeted bronchus, the tracheal cuff will be inflated and ventilation of the lungs started. Fiberoptic bronchoscopic assessment of adequate bronchial cuff placement will be followed by DLT placement. DLT insertion time will be defined as from the time the laryngoscope passed the patient's lips until three complete end-tidal carbon dioxide cycles were displayed on the monitor. Intubation success rate at the first attempt will be recorded by the same observer. The difficulty of DLT insertion and delivery will be assessed by the operator, using NRS ranging from 0 to 10. The NRS results will be grouped as 0 = none, 1-3 = mild, 4-6 = moderate, and 7-10 = severe. C/L degrees were classified as four degrees (I, IIA, IIB, and III) and will be assessed by the same operator. If the degree will be not class I, external laryngeal pressure will be provided by an assistant. Time required to successful intubation. Intubation time is defined as the time taken for insertion of the blade between the teeth till the tracheal tube cuffٴ passed through the vocal cords. Failure of intubation was defined as any intubation attempt of >120 s or inability to intubate. Number of intubation attempts, Ease of laryngoscope insertion, Quality of view by Cormack and Lehane grade . Assist maneuvers. Intubation difficult score indicates the degree of difficulty of intubation using 7 parameters (0=easy intubation, 0 ˂IDS≤5 =slight difficulty, 5 < IDS =moderate to major diffculty, IDS= ∞ impossible intubation) . The time taken for fiberoptic bronchoscopy was defined as the time from endobronchial intubation to placement confirmation using fiberoptic bronchoscopy. The operators examined blade surfaces for blood after removal. Hemodynamic parameters (mean arterial blood pressure and heart rate) will be recorded 10 min before induction and 1, 3, and 5 min after intubation. After the assessment by fiberoptic bronchoscopy, the oral cavity, pharynx, larynx and teeth will be examined for signs of laceration or bleeding by an independent investigator who will be unaware of the type of laryngoscope used. One day after surgery, an independent investigator will interview patients to assess the presence of sore throat and hoarseness of voice.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* BMI < 35 kg/m2
* Mallampati score of 1 or 2

Exclusion Criteria:

* Patients with risk of gastric aspiration
* Patients with risk of gastric aspiration
* Presence of any predictors of difficult intubation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Double lumen tube insertion times in seconds | 2 minutes
  Double lumen tube insertion times by the three types of laryngoscopes were recorded
first-pass success rates | 2 minutes
  Double lumen tube insertion first-pass success ratesby the three types of laryngoscopes were recorded

SECONDARY OUTCOMES:
Blood pressure measurement in mm Hg | 150 minutes
  During intubation and then every 15 minutes in mm Hg
Heart rate measurement in beat/minute | 150 minutes
  During intubation and then every 15 minutes in beat/minute

CONTACTS AND LOCATIONS:
Locations (1):
- Mona Mohamed Mogahed, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided